CLINICAL TRIAL: NCT03629873
Title: A Phase 2 Study Evaluating Efficacy and Safety of Chi-BEAC Combining With Auto-HSCT to Treat Aggressive Lymphoma Subjects
Brief Title: Efficacy and Safety of Chi-BEAC Combining With Auto-HSCT to Treat Aggressive Lymphoma Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-Chi-BEAC-HSCT
Record Dates: First submitted 2018-08-05; First posted 2018-08-14 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Mantle Cell Lymphoma; Peripheral T Cell Lymphoma; Double-hit Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell; Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Carmustine; Etoposide; Cytarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chidamide — Chidamide 30mg po d-7、-4、0、3; Carmustine 300mg/m^2 IVD d-6; Etoposide 150mg/m^2/d qd IVD d-5~-2; Cytarabine 150mg/m^2 q12h IVD d-5~-2; Cyclophosphamide 1.0g/m^2/d qd IVD d-5~-2
  Other Names: Carmustine; Etoposide; Cytarabine; Cyclophosphamide; Autologous hematopoeitic stem cell transplantation

SUMMARY:
This is a single arm, multi-center, open study to evaluating efficacy and safety of Chi-BEAC combining with auto-HSCT to treat aggressive lymphoma Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Aggressive lymphoma subjects: diffuse large B cell lymphoma confirmed by immunohistochemistry, aaIPI≥2 or double-hit lymphoma, as first-line consolidation; diffuse large B cell lymphoma as second-line consolidation therapy; peripheral T-cell lymphoma except ALK-positive type, as first-line or second-line consolidation therapy; mantle cell lymphoma, as first-line or second-line consolidation therapy.
2. Adequate organ system function including:

   Creatinine clearance rate ≥ 80ml/min and creatinine < 160μmol/L ALT/AST ≤ 2 upper limit of normal Total Bilirubin < 2 upper limit of normal FEV1、FVC and DLCO ≥ 50% predictive value Left ventricular ejection fraction ≥ 50% No Symptomatic arrhythmia
3. Age 18-60 years, male and female
4. ECOG score 0-1
5. Number of neutrophil ≥ 1.5×10^9/L, number of platelet ≥ 70×10^9/L, concentration of hemoglobin ≥ 90g/L, number of CD34+ cells ≥ 2.0×10^6/kg
6. Expected survival ≥ 12 weeks
7. Volunteered to participate in this study and signed informed consent

Exclusion Criteria:

1. Have evidence of CNS lymphoma
2. Relapse after autologous hematopoietic stem cell transplantation
3. Active hepatitis B or hepatitis C virus infection
4. Severe active infection
5. HIV-infected persons
6. Liver cirrhosis or hepatic fibrosis
7. QTc > 500ms
8. Have mental disorder or unable to sign informed consent
9. History of drug abuse and intemperance
10. Women who are pregnant or lactating or have breeding intent
11. The investigators believe that any increase in the risk of the subject or interference with the results of the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 2 years after transplantation

SECONDARY OUTCOMES:
Overall survival | 2 years after transplantation
Complete remission | 3 months after transplantation
Time of hematopoietic reconstitution | 15 days, 1 month
Non-relapse mortality | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China